CLINICAL TRIAL: NCT02199691
Title: A Phase II Study of the Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Healthy Adolescents
Brief Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Healthy Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MET50; U1111-1143-8537 (Other: WHO)
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; MenACYW Conjugate vaccine; MENVEO vaccine; Adacel®; GARDASIL®
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines; adacel; Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal-vaccine naïve participants aged 10 to 17 years received a single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W135) Tetanus Toxoid Conjugate Vaccine
- Group 2: MENVEO® Vaccine (Active Comparator): Healthy, meningococcal-vaccine naïve participants aged 10 to 17 years received a single dose of MENVEO® vaccine on Day 0.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine
- Group 3: MenACYW Conjugate Vaccine+Tdap+HPV (Experimental): Healthy, meningococcal-vaccine naïve participants aged 10 to 17 years received a single dose of MenACYW Conjugate vaccine, Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Tdap), and Dose 1 of HPV Vaccine on Day 0. HPV Vaccine Dose 2 and Dose 3 were given at 2 and 6 months, respectively, after Dose 1 given on Day 0.
  Interventions: Biological: Adacel®: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed; Biological: GARDASIL®: Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant; Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W135) Tetanus Toxoid Conjugate Vaccine
- Group 4: Tdap+HPV (Active Comparator): Healthy, meningococcal-vaccine naïve participants aged 10 to 17 years received a single dose of Tdap and Dose 1 of HPV Vaccine on Day 0. HPV Vaccine Dose 2 and Dose 3 were given at 2 and 6 months, respectively, after Dose 1 given on Day 0.
  Interventions: Biological: Adacel®: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed; Biological: GARDASIL®: Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W135) Tetanus Toxoid Conjugate Vaccine — 0.5 milliliter (mL), Intramuscular (IM)
  Other Names: MenACYW Conjugate vaccine
  Arms: Group 1: MenACYW Conjugate Vaccine
Biological: Meningococcal (Groups A, C, Y and W135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine — 0.5 mL, IM
  Other Names: MENVEO®
  Arms: Group 2: MENVEO® Vaccine
Biological: Adacel®: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed — 0.5 mL, IM
  Other Names: Adacel® (Tdap)
  Arms: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV
Biological: GARDASIL®: Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant — 0.5 mL, IM
  Other Names: GARDASIL® (HPV)
  Arms: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W135) Tetanus Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular (IM)
  Other Names: MenACYW Conjugate vaccine
  Arms: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV
Biological: Adacel®: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed — 0.5 mL, IM
  Other Names: Adacel® (Tdap)
  Arms: Group 4: Tdap+HPV
Biological: GARDASIL®: Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant — 0.5 mL, IM
  Other Names: GARDASIL® (HPV)
  Arms: Group 4: Tdap+HPV

SUMMARY:
The purpose of the study was to evaluate the immunogenicity and describe the safety of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine compared to the licensed vaccine MENVEO® in adolescents 10 to 17 years of age in the United States (US). This study also evaluated the immunogenicity and safety of MenACYW Conjugate vaccine when given alone compared to when given concomitantly with tetanus, diphtheria, acellular pertussis (Tdap) vaccine and human papilloma virus (HPV) vaccine.

Primary objective:

* To evaluate the antibody responses to the antigens present in MenACYW Conjugate vaccine when MenACYW Conjugate vaccine was given alone compared to those when MENVEO vaccine was given alone.

Secondary objective:

* To evaluate the antibody responses to the antigens present in MenACYW Conjugate vaccine, when MenACYW Conjugate vaccine was given concomitantly with Tdap and HPV vaccines, compared to those when it was given alone.
* To evaluate the antibody responses to the antigens present in Tdap vaccine, when Tdap vaccine was given concomitantly with MenACYW Conjugate vaccine and HPV vaccine, compared to those when Tdap vaccine was given with HPV vaccine only.
* To evaluate the antibody responses to the antigens present in HPV vaccine after the 3-dose series, when the first dose of HPV vaccine is given concomitantly with MenACYW Conjugate vaccine and Tdap vaccine, compared to those when the first dose of HPV vaccine is given with Tdap vaccine only.

Observational objective:

* To describe the safety profile of MenACYW Conjugate vaccine, compared to that of the licensed vaccine MENVEO®, and when MenACYW Conjugate vaccine was given with Tdap and HPV vaccines.

DETAILED DESCRIPTION:
Healthy adolescents were randomized and received a single dose of their assigned vaccines. They were assessed for immunogenicity at baseline (pre-vaccination) and at 30 days post-vaccination. Safety information were collected post-vaccination and throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 17 years on the day of inclusion.
* Informed consent form was signed and dated by the parent(s) or another legally acceptable representative.
* Assent form was signed and dated by the participant.
* Participant and parent legally acceptable representative were able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination).
* Participation in the 4 weeks preceding the first trial vaccination(s) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination(s) or planned receipt of any vaccine in the 4 weeks prior to or following any trial vaccination except for influenza vaccination, which may be received at least 2 weeks before or after any study vaccines. This exception included monovalent influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or any mono- or polyvalent polysaccharide or conjugate meningococcal vaccine containing A, C, W, or Y antigens.
* History of vaccination with any tetanus, diphtheria, or pertussis vaccine within the previous 4 years.
* Previous human papilloma virus (HPV) vaccination.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (i.e., participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances, including encephalopathy (e.g., coma, decreased level of consciousness, prolonged seizures) within 7 days of administration of a previous pertussis antigen-containing vaccine.
* Personal history of Guillain-Barré syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within at least 10 years of the proposed study vaccination.
* Verbal report of thrombocytopenia, contraindicating intramuscular vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness (e.g., human immunodeficiency virus [HIV] hepatitis B, hepatitis C) that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >= 100.4 degree fahrenheit [°F]). A prospective participant was not included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1715 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2015-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (32):
- United States (31):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Downey, California
  - San Diego, California
  - Miami Beach, Florida
  - Wichita, Kansas
  - Bardstown, Kentucky
  - Nicholasville, Kentucky
  - Columbia, Maryland
  - Lincoln, Nebraska
  - Cleveland, Ohio
  - Dayton, Ohio
  - Norman, Oklahoma
  - Erie, Pennsylvania
  - Charleston, South Carolina
  - Kingsport, Tennessee
  - Tullahoma, Tennessee
  - Layton, Utah
  - Orem, Utah
  - Payson, Utah
  - Provo, Utah
  - Roy, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Spanish Fork, Utah
  - Syracuse, Utah
  - West Haven, Utah
  - West Jordan, Utah
  - Charlottesville, Virginia
  - Midlothian, Virginia
  - Spokane, Washington
- San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Chang LJ, Hedrick J, Christensen S, Pan J, Jordanov E, Dhingra MS. A Phase II, randomized, immunogenicity and safety study of a quadrivalent meningococcal conjugate vaccine, MenACYW-TT, in healthy adolescents in the United States. Vaccine. 2020 Apr 23;38(19):3560-3569. doi: 10.1016/j.vaccine.2020.03.017. Epub 2020 Mar 21. PMID 32209248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 40 centers in the Unites States (US) from 22 July 2014 to 25 February 2015.
Pre-assignment Details: A total of 1715 participants were enrolled and randomized in the study.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy, meningococcal-vaccine naïve participants aged 10 to 17 years received a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine on Day 0.
- Group 3: MenACYW Conjugate Vaccine+Tdap+HPV: Healthy, meningococcal-vaccine naïve participants aged 10 to 17 years received a single dose of MenACYW Conjugate vaccine, Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Tdap), and Dose 1 of Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant (HPV) on Day 0. HPV Vaccine Dose 2 and Dose 3 were given at 2 and 6 months, respectively, after Dose 1 given on Day 0.
- Group 4: Tdap+HPV: Healthy, meningococcal-vaccine naïve participants aged 10 to 17 years received a single dose of Tdap and Dose 1 of HPV on Day 0. HPV Vaccine Dose 2 and Dose 3 were given at 2 and 6 months, respectively, after Dose 1 given on Day 0.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV | Group 4: Tdap+HPV
Started | 505 | 507 | 403 | 300
Safety Analysis Set (SafAS) (SafAS:participants who received at least 1 dose of study vaccine(s) & had any safety data available.) | 503 | 501 | 392 | 296
Completed | 495 | 500 | 376 | 270
Not Completed | 10 | 7 | 27 | 30
Not completed — Protocol Violation | 3 | 3 | 6 | 7
Not completed — Withdrawal by Subject | 5 | 3 | 12 | 13
Not completed — Lost to Follow-up | 2 | 1 | 9 | 10

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV | Group 4: Tdap+HPV | Total
Number analyzed (Participants) | 505 | 507 | 403 | 300 | 1715
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (1.39) | 11.4 (1.39) | 11.3 (1.06) | 11.4 (1.41) | 11.4 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 232 | 197 | 144 | 832
  Male | 246 | 275 | 206 | 156 | 883
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 4 | 1 | 8
  Asian | 3 | 3 | 1 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 2 | 5 | 10
  Black or African American | 30 | 22 | 15 | 18 | 85
  White | 442 | 456 | 361 | 261 | 1520
  More than one race | 26 | 24 | 20 | 12 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 505 | 507 | 403 | 300 | 1715

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Vaccine Seroresponse Measured by Serum Bactericidal Assay Using Human Complement (hSBA) Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With Either MenACYW Conjugate Vaccine or MENVEO® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA. The hSBA vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers greater than or equal to (>=) 1:8 for participants with pre-vaccination hSBA titers less than (<) 1:8 or at least a 4-fold increase in hSBA titers from pre- to post vaccination for participants with pre-vaccination hSBA titers >= 1:8. Data for this outcome measure was not planned to be collected and analyzed for Group 4:Tdap+HPV.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on Per-Protocol Analysis Set-1(PPAS-1) defined for accessing the ACYW & Tdap immune response data for all participants after they had received vaccination(s) at Visit 1(Day 0) & completed blood sampling (BL) at Visit 2(Day 30). Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Number analyzed (Participants) | 463 | 464
percentage of participants
  Serogroup A | 75.6 [71.4 to 79.4] | 66.4 [61.9 to 70.7]
  Serogroup C: number analyzed (Participants) | 462 | 463
  Serogroup C | 97.2 [95.2 to 98.5] | 72.6 [68.3 to 76.6]
  Serogroup Y: number analyzed (Participants) | 462 | 464
  Serogroup Y | 97.0 [95.0 to 98.3] | 80.8 [76.9 to 84.3]
  Serogroup W | 86.2 [82.7 to 89.2] | 66.6 [62.1 to 70.9]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup A; Test type: Non-Inferiority — 95% confidence interval (CI) of the difference was calculated from the Wilson Score Method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference between the 2 percentages was > -10%; Percentage Difference = 9.2, 95% CI 2-sided [3.4 to 15]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup C; Test type: Non-Inferiority — 95% CI of the difference was calculated from the Wilson Score Method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference between the 2 percentages was > -10%; Percentage Difference = 24.6, 95% CI 2-sided [20.3 to 29]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = 16.2, 95% CI 2-sided [12.3 to 20.2]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = 19.6, 95% CI 2-sided [14.2 to 24.8]

2. Secondary Outcome: Percentage of Participants Achieving hSBA Vaccine Seroresponse Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With Either MenACYW Conjugate Vaccine or MenACYW Conjugate Vaccine Given With Tdap and HPV Vaccines
Description: Antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA. The hSBA vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >= 1:8 for participants with pre-vaccination hSBA titers < 1:8 or at least a 4-fold increase in hSBA titers from pre- to post vaccination for participants with pre-vaccination hSBA titers >= 1:8.
Time Frame: Day 30 (post-vaccination on Day 0)
Population: Analysis was performed on PPAS-1. Here 'Number analyzed' signifies number of participants with available data for specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 4: Tdap+HPV.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV
Number analyzed (Participants) | 463 | 360
percentage of participants
  Serogroup A | 75.6 | 80.6
  Serogroup C: number analyzed (Participants) | 462 | 360
  Serogroup C | 97.2 | 97.2
  Serogroup Y: number analyzed (Participants) | 462 | 360
  Serogroup Y | 97.0 | 95.6
  Serogroup W | 86.2 | 83.9
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: MenACYW Conjugate Vaccine+Tdap+HPV; Serogroup A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = 5, 95% CI 2-sided [-0.8 to 10.5]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: MenACYW Conjugate Vaccine+Tdap+HPV; Serogroup C; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = 0, 95% CI 2-sided [-2.5 to 2.4]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: MenACYW Conjugate Vaccine+Tdap+HPV; Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = -1.4, 95% CI 2-sided [-4.3 to 1.2]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: MenACYW Conjugate Vaccine+Tdap+HPV; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = -2.3, 95% CI 2-sided [-7.3 to 2.6]

3. Secondary Outcome: Geometric Mean Concentrations (GMCs) of PT, FHA, PRN, and FIM Antibodies Following Vaccination With Either MenACYW Conjugate Vaccine Given With Tdap and HPV Vaccines or Tdap and HPV Vaccines
Description: Anti-Pertussis toxoid (PT), Filamentous hemagglutinin (FHA), Pertactin (PRN), and Fimbriae types 2 and 3 (FIM) antibodies were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 30 (post-vaccination on Day 0)
Population: Analysis was performed on PPAS-1. Here 'Number analyzed' signifies number of participants with available data for specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 1: MenACYW Conjugate vaccine and Group 2: MENVEO® vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units (EU)/mL
Arm/Group | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV | Group 4: Tdap+HPV
Number analyzed (Participants) | 360 | 263
ELISA units (EU)/mL
  Anti-Pertussis toxoid (PT): number analyzed (Participants) | 339 | 258
  Anti-Pertussis toxoid (PT) | 37.5 [33.8 to 41.7] | 44.4 [39.5 to 49.9]
  Filamentous hemagglutinin (FHA): number analyzed (Participants) | 358 | 263
  Filamentous hemagglutinin (FHA) | 180 [168 to 194] | 242 [218 to 268]
  Pertactin (PRN) | 200 [177 to 225] | 265 [231 to 304]
  Fimbriae types 2 and 3 (FIM): number analyzed (Participants) | 350 | 262
  Fimbriae types 2 and 3 (FIM) | 339 [285 to 403] | 499 [414 to 601]
Statistical Analysis 1: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; PT: Geometric Mean Ratio; Test type: Non-Inferiority — 95% CI of the difference was calculated from the Wilson Score Method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the ratio was >2/3; Geometric Mean Ratio = 0.845, 95% CI 2-sided [0.722 to 0.99]
Statistical Analysis 2: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; FHA: Geometric Mean Ratio; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Geometric Mean Ratio = 0.746, 95% CI 2-sided [0.661 to 0.842]
Statistical Analysis 3: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; PRN: Geometric Mean Ratio; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Geometric Mean Ratio = 0.753, 95% CI 2-sided [0.627 to 0.903]
Statistical Analysis 4: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; FIM: Geometric Mean Ratio; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Geometric Mean Ratio = 0.679, 95% CI 2-sided [0.525 to 0.878]

4. Secondary Outcome: Percentage of Participants Achieving Anti-Tetanus and Anti-Diphtheria Concentrations >= 1.0 International Unit (IU)/mL Following Vaccination With Either MenACYW Conjugate Vaccine Given With Tdap and HPV Vaccines or Tdap and HPV Vaccines
Description: Anti-Diphtheria antibodies were measured by a toxin neutralization test. Anti-Tetanus antibodies were measured by ELISA.
Time Frame: Day 30 (post-vaccination on Day 0)
Population: Analysis was performed on PPAS-1. Here "Number analyzed' signifies number of participants with available data for specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 1: MenACYW Conjugate vaccine and Group 2: MENVEO® vaccine.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV | Group 4: Tdap+HPV
Number analyzed (Participants) | 360 | 263
percentage of participants
  Diphtheria | 97.8 [95.7 to 99.0] | 98.9 [96.7 to 99.8]
  Tetanus: number analyzed (Participants) | 360 | 262
  Tetanus | 99.7 [98.5 to 100.0] | 99.6 [97.9 to 100.0]
Statistical Analysis 1: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; Serogroup Diphtheria; Test type: Non-Inferiority — 95% CI of the difference was calculated from the Wilson Score Method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference between the 2 percentages was >-10%; Percentage Difference = -1.1, 95% CI 2-sided [-3.3 to 1.3]
Statistical Analysis 2: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; Serogroup Tetanus; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Percentage Difference = 0.1, 95% CI 2-sided [-1.2 to 1.9]

5. Secondary Outcome: Percentage of Participants Achieving Seroconversion for Anti-HPV6, HPV11, HPV16, and HPV18 Antibodies Following Vaccination With Either MenACYW Conjugate Vaccine Given With Tdap and HPV Vaccines or Tdap and HPV Vaccines
Description: Anti-HPV 6, 11, 16, and 18 antibodies were measured using a competitive Luminex immunoassay. Seroconversion was defined as changing serostatus from seronegative to seropositive. Cutoff values for HPV seropositivity were >= 20 milli-Merck units per milliliter (mMU/mL) for types 6 and 16, >= 16 mMU/mL for type 11, and >= 24mMU/mL for type 18.
Time Frame: Day 210 (post-vaccination on Day 0)
Population: Per-Protocol Analysis Set-2(PPAS-2)defined for accessing HPV immune response data for participants in Group 3 & 4 after they received third HPV vaccination at Visit 4(Day 180)& completed blood sample at Visit 5(BL3 [Day 210]).Data for this outcome measure was not planned to be collected and analyzed for Groups 1 and 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV | Group 4: Tdap+HPV
Number analyzed (Participants) | 242 | 164
percentage of participants
  HPV Type 6 | 97.5 [94.7 to 99.1] | 95.7 [91.4 to 98.3]
  HPV Type 11 | 99.6 [97.7 to 100.0] | 98.8 [95.7 to 99.9]
  HPV Type 16 | 99.2 [97.0 to 99.9] | 98.8 [95.7 to 99.9]
  HPV Type 18 | 99.2 [97.0 to 99.9] | 98.8 [95.7 to 99.9]
Statistical Analysis 1: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; HPV Type 6; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Percentage Difference = 1.8, 95% CI 2-sided [-1.8 to 6.3]
Statistical Analysis 2: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; HPV Type 11; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Percentage Difference = 0.8, 95% CI 2-sided [-1.3 to 3.9]
Statistical Analysis 3: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; HPV Type 16; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Percentage Difference = 0.4, 95% CI 2-sided [-1.9 to 3.6]
Statistical Analysis 4: Comparison: Group 3: MenACYW Conjugate Vaccine+Tdap+HPV vs Group 4: Tdap+HPV; HPV Type 18; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Percentage Difference = 0.4, 95% CI 2-sided [-1.9 to 3.6]

6. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions (Pain, Erythema, Swelling) Following Vaccination With MenACYW Conjugate Vaccine or MENVEO® Vaccine at Day 0: Group 1 and Group 2
Description: A Solicited Reaction (SR) was an Adverse Event (AE) that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). Solicited injection site reactions included: Pain, Erythema, and Swelling.
Time Frame: Within 7 days after vaccines injections at Day 0
Population: Analysis was performed on Safety Analysis Set (SafAS) defined as participants who received at least one dose of the study vaccine(s) and had any safety data available. All participants had their safety data analyzed according to vaccine(s) they actually received. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Number analyzed (Participants) | 503 | 501
Participants
  Pain: number analyzed (Participants) | 496 | 492
  Pain | 224 | 209
  Erythema: number analyzed (Participants) | 496 | 491
  Erythema | 25 | 37
  Swelling: number analyzed (Participants) | 496 | 491
  Swelling | 27 | 32

7. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions (Pain, Erythema, Swelling) Following Vaccination With MenACYW Conjugate Vaccine Given With Tdap and HPV Vaccines at Day 0: Group 3
Description: A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). Solicited injection site reactions included: Pain, Erythema, and Swelling.
Time Frame: Within 7 days after vaccines injections at Day 0
Population: Analysis was performed on SafAS. Here "Overall number of participants analyzed" = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV
Number analyzed (Participants) | 388
Participants
  MenACYW site: Pain | 183
  MenACYW site: Erythema | 15
  MenACYW site: Swelling | 17
  Tdap site: Pain | 286
  Tdap site: Erythema | 28
  Tdap site: Swelling | 24
  HPV site: Pain | 288
  HPV site: Erythema | 31
  HPV site: Swelling | 26

8. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions (Pain, Erythema, Swelling) Following Vaccination With Tdap and HPV Vaccines at Day 0: Group 4
Description: as for outcome 7
Time Frame: Within 7 days after vaccines injections at Day 0
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Tdap+HPV
Number analyzed (Participants) | 289
Participants
  Tdap site: Pain | 211
  Tdap site: Erythema | 14
  Tdap site: Swelling | 20
  HPV site: Pain | 201
  HPV site: Erythema | 16
  HPV site: Swelling | 23

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to 30 days after last vaccination. SR data were collected within 7 days after any vaccination. Serious adverse events (SAEs) data were collected throughout the study (up to 180 days after vaccination for Group 1 and 2, and up to 210 days after vaccination on Day 0 for Group 3 and 4).
Description: Analysis was performed on Safety Analysis Set. A SR was an AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV | Group 4: Tdap+HPV
All-Cause Mortality (participants affected / at risk) | 0/503 | 0/501 | 0/392 | 0/296
Serious Adverse Events (participants affected / at risk) | 4/503 | 4/501 | 4/392 | 4/296
Other Adverse Events (participants affected / at risk) | 331/503 | 337/501 | 348/392 | 263/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=503) | Group 2: MENVEO® Vaccine (N=501) | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV (N=392) | Group 4: Tdap+HPV (N=296)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Staphylococcal Scalded Skin Syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abnormal Behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=503) | Group 2: MENVEO® Vaccine (N=501) | Group 3: MenACYW Conjugate Vaccine+Tdap+HPV (N=392) | Group 4: Tdap+HPV (N=296)
Injection Site Erythema (General disorders) | 25 (25) | 37 (37) | 44 (74) | 24 (30)
Injection Site Pain (General disorders) | 224 (224) | 209 (209) | 327 (759) | 234 (412)
Injection Site Swelling (General disorders) | 27 (27) | 32 (32) | 42 (67) | 32 (43)
Malaise (General disorders) | 130 (130) | 131 (131) | 113 (113) | 81 (81)
Pharyngitis (Infections and infestations) | 15 (15) | 32 (34) | 22 (22) | 14 (16)
Upper Respiratory Tract Infection (Infections and infestations) | 24 (27) | 30 (33) | 27 (31) | 12 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 175 (175) | 173 (173) | 239 (239) | 161 (161)
Headache (Nervous system disorders) | 155 (165) | 159 (168) | 137 (145) | 87 (89)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.